CLINICAL TRIAL: NCT06045676
Title: Electrocardiographic Changes Among Epileptic and Non Epileptic Seizures in Children at Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amany Khalaf Allah Elzanaty, Resident, Sohag University
Other Study IDs: Soh-Med-23-09-06MS
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Seizures
MeSH Terms: conditions — Seizures | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Drug Resistant Epilepsy: Seizures Not Respond to two lines of Anti epileptic Medications
  Interventions: Device: ECG
- Drug Responsive Epilepsy: Seizures Respond to one or two lines of Anti epileptic Medications
  Interventions: Device: ECG
- Febrile Seizures: type of seizure occurring due to fever over 38 °C without a history of convulsion
  Interventions: Device: ECG
- Breath Holding Spells: children's behaviors look like epileptic seizures due to crying up to a minute followed by losing consciousness
  Interventions: Device: ECG
- Control: Healthy Children free from any convulsion
  Interventions: Device: ECG

INTERVENTIONS:
Device: ECG — ECG with special comment on QT interval. QT interval was measured as the distance from the beginning of the Q wave to the end of the T wave at least in eight leads from the standard ECG.

SUMMARY:
Epilepsy is a chronic disease triggered by increased impulsiveness of nerve cells in the brain and may require a lifelong treatment. Epilepsy is confirmed by two or more unprovoked seizures in more than 24 hours. Febrile Convulsion is another type of seizure occurring due to fever over 38 °C without a history of convulsion, CNS infection, electrolyte imbalance, metabolic disorder, intoxication, and trauma. Unlike epileptic seizures, there are non-epileptic seizures such as Breath Holding Spells that affect children's behaviors and often look like epileptic seizures.

QT parameters elongation show the danger of dysrhythmia and unexpected sicknesses such as cardiomyopathy, mitral valve prolapse, ischemic coronary illness, and kidney disorders.

Many investigators have reported changes in QT parameters in various diseases such as diabetes mellitus, celiac disease, thalassemia , epilepsy ,Breath holding spells and febrile seizure.

ELIGIBILITY:
Inclusion Criteria:

* children with drug resistant epilepsy.
* febrile seizures.
* age of 1 year to 12 years.

Exclusion Criteria:

* age below 1 year and above 12 years
* children with convulsion secondary cns infection , encephalitis, encephalopathy , toxic and metabolic problem

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with drug resistant epilepsy , responsive epilepsy , febrile seizures and breath holding spells with age of 1 year to 12 years
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-09-25 (Estimated); Primary Completion 2024-09-25 (Estimated); Study Completion 2024-09-25 (Estimated)

PRIMARY OUTCOMES:
QT interval | 12 months
  Distance from the beginning of the Q wave to the end of the T wave at least in eight leads from the standard ECG

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided